CLINICAL TRIAL: NCT01993615
Title: A Supervised Physical Therapy Program vs. Arthroscopic Surgery for Femoroacetabular Impingement: A Randomized Clinical Trial
Brief Title: A Physical Therapy Program Versus Surgery for Femoroacetabular Impingement: Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dan Rhon, Director of Physical Therapy, Department of PM&R, Madigan Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 213011
Record Dates: First submitted 2013-10-30; First posted 2013-11-25 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-07

CONDITIONS: Femoroacetabular Impingement
Keywords: FAI; femoroacetabular impingement; hip pain; hip arthroscopy; physical therapy
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Arthroscopy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arthroscopic Surgery (Active Comparator): Arthroscopic surgery at the femoroacetabular joint, followed by a standardized post-operative rehabilitation protocol in physical therapy.
  Interventions: Procedure: Arthroscopic Surgery
- Physical Therapy (Active Comparator): An impairment-based supervised in-clinic physical therapy program.
  Interventions: Procedure: Physical Therapy

INTERVENTIONS:
Procedure: Arthroscopic Surgery — The hip arthroscopy will consist of acetabular rim trimming, labral repair or debridement and femoroplasty, all as indicated based on the surgeon's clinical judgment with input from pre-operative imaging, exam findings and intra-operative findings.
  Arms: Arthroscopic Surgery
Procedure: Physical Therapy — Subjects will participate in two 45-minute sessions for six weeks (total of 12 sessions). The physical therapy treatment plan will be based on individual impairments identified during the initial evaluation, and include manual therapy to the hip, lumbar spine, and pelvis, as well as therapeutic exercise all tailored to individual patient impairments.
  Arms: Physical Therapy

SUMMARY:
The purpose of this study is to compare the outcomes for patients that receive two different treatments used for FAI (Femoroacetabular Impingement). The programs are 1) a 6-week supervised physical therapy program and 2) arthroscopic surgery. Enrollment is limited to patients that have already been determined surgical candidates. The study is following patients for a 2-year period.

DETAILED DESCRIPTION:
This study plans to enroll a total of 60 Tricare beneficiaries primarily from the Madigan Healthcare System with a diagnosis of FAI that are surgical candidates and have already failed at least six weeks of conservative treatment.

This is a randomized controlled study comparing outcomes for the standard treatment for FAI and/or acetabular labral pathology (arthroscopy with or without labral repair) versus physical therapy. For subjects in the arthroscopy group, the surgery will be performed by the Orthopedic Surgical Service at Madigan Army Medical Center.

Subjects randomized to the physical therapy group will follow a treatment plan implemented by a physical therapist within the Madigan Army Healthcare System.

After consent, subjects will be randomized into one of two arms (Group I = hip arthroscopy, Group II = physical therapy). Group I will undergo hip arthroscopy with or without labral repair. Group II will follow a FAI-based physical therapy program x 12 sessions (6 weeks).

The arthroscopy group will complete outcome measures at time of consent and following surgery at 6 months, 1 year and 2 year time periods. Subjects in this group will follow a standardized post-operative rehabilitation protocol.

The physical therapy group will complete outcomes measures at time of consent and at 6 month, 1 year and 2 year time periods following the initial physical therapy evaluation. Subjects in this group will complete 6 weeks of an impairment-based physical therapy program.

In addition to the outcome measures taken, healthcare utilization and associated costs for hip-related care during this 2-year period will also calculated for comparison between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Tricare beneficiaries between the ages of 18 and 65
* Diagnosis of FAI and/or labral pathology confirmed by a combination of the following:

  * Pain at the anterior hip or groin
  * Pain with hip flexion
  * Positive FADIR test
  * Patient report relief of pain after intra-articular injection
* Surgical candidate for hip arthroscopy defined by (must have both):

  * No less than 2 mm of joint space based on imaging (CT scan, radiographs and MR arthrogram)
  * Positive crossover sign and/or alpha angle >50 deg based on imaging (CT scan, radiographs and MR arthrogram)
* Failed 6 weeks of conservative management

Exclusion Criteria:

* Pregnancy
* Has other concurrent systemic disease that may affect the condition (cancer, rheumatoid arthritis, or other systemic arthralgia/arthritis)
* Has had surgery on the same hip that will be analyzed in the study
* Diagnosis of hip osteoarthritis is more likely
* Clearing the lumbar spine reproduces the patient's hip symptoms
* Plans to move/relocate out of the local area within 6 months
* Pending litigation for their hip condition
* Unable to give informed consent to participate in the study
* Unable to speak or read or write in English (due to inability to fill out outcome measures)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Mansell, PT, DPT, Principal Investigator — Madigan Army Medical Center; Daniel Rhon, DPT, DSc, Study Chair — Madigan Army Medical Center
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data sharing must go through a Data Sharing Agreement approved by the US Defense Health Agency

REFERENCES:
- [Derived] Mansell NS, Rhon DI, Meyer J, Slevin JM, Marchant BG. Arthroscopic Surgery or Physical Therapy for Patients With Femoroacetabular Impingement Syndrome: A Randomized Controlled Trial With 2-Year Follow-up. Am J Sports Med. 2018 May;46(6):1306-1314. doi: 10.1177/0363546517751912. Epub 2018 Feb 14. PMID 29443538
- [Derived] Mansell NS, Rhon DI, Marchant BG, Slevin JM, Meyer JL. Two-year outcomes after arthroscopic surgery compared to physical therapy for femoracetabular impingement: A protocol for a randomized clinical trial. BMC Musculoskelet Disord. 2016 Feb 4;17:60. doi: 10.1186/s12891-016-0914-1. PMID 26846934

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from the orthopaedic clinic at Madigan Army Medical Center
Period: Overall Study
Arm/Group | Arthroscopic Surgery | Physical Therapy
Started | 40 | 40
Completed | 39 | 40
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arthroscopic Surgery | Physical Therapy | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (7.4) | 30.6 (7.4) | 30.1 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 21 | 26 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 5 | 4 | 9
  White | 30 | 28 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Hip Outcome Score - ADL Subscale at 24 Months
Description: The Hip Outcome Score is designed to assess higher-level activities (i.e. those required in athletics) and has demonstrated validity in a study of patients at a mean of three years following hip arthroscopy. Additionally, a 2011 study states that the HOS has the greatest amount of clinimetric evidence (rigor of rating scales and indexes for the description of clinical phenomena). Only three published patient-reported outcome instruments utilized to assess FAI and labral pathology use clinimetric evidence and the HOS was identified as the most proven instrument. The HOS ADL Subscale consisted of 19 questions, each scored on a 5-point scale from 0 (unable to do) to 4 (no difficulty). The final score is calculated by taking the raw score, dividing it by the number of total questions answered multipled by 4 x 100 for a final score that ranges from 0 to 100%, with lower scores associated with greater limitation in Activities of Daily Living (ADL).
Time Frame: 24 months
Population: Intention to treat analysis including only participants that received any treatment (6 participants that were enrolled never returned for treatment)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arthroscopic Surgery | Physical Therapy
Number analyzed (Participants) | 37 | 37
score on a scale | 69.3 [62.5 to 76.2] | 73.1 [66.1 to 80.3]

2. Primary Outcome: Hip Outcome Score - Sport Subscale at 24 Months
Description: The Hip Outcome Score is designed to assess higher level activities (i.e. those required in athletics) and has demonstrated validity in a study of patients at a mean of three years following hip arthroscopy. Additionally, a 2011 study states that the HOS has the greatest amount of clinimetric evidence (rigor of rating scales and indexes for the description of clinical phenomena). Only three published patient-reported outcome instruments utilized to assess FAI and labral pathology use clinimetric evidence and the HOS was identified as the most proven instrument. The HOS Sport Subscale consists of 9 questions, each scored on a 5-point scale from 0 (unable to do) to 4 (no difficulty). The final score is calculated by taking the raw score, dividing it by the number of total questions answered multipled by 4 x 100 for a final score that ranges from 0 to 100%, with lower scores associated with greater limitations in Sports-related activities.
Time Frame: 24 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arthroscopic Surgery | Physical Therapy
Number analyzed (Participants) | 37 | 37
score on a scale | 55.3 [46.2 to 64.4] | 57.1 [47.8 to 66.3]

3. Secondary Outcome: Group Differences in International Hip Outcome Score (IHOT33) to 24 Months
Description: The iHOT33 is a quality-of-life patient-reported outcome measure that uses a visual analog scale response format for young, active patients with hip pathology. This 33-item questionnaire includes four sections: symptoms and functional limitations, sports and recreational activities, job related concerns and social, emotional and lifestyle concerns. This outcome measure has shown to be reliable; shows face, content and contrast validity and is highly responsive to clinical change. It uses a visual analog scale with the verbal anchors "no problems at all" on the far right and "significantly impaired" on the left. The total score is calculated as a simple mean of the responses ranging from 0 to 100, with 100 representing the best possible quality-of-life score.
Time Frame: 24 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arthroscopic Surgery | Physical Therapy
Number analyzed (Participants) | 37 | 37
score on a scale | 51.2 [42.5 to 59.9] | 44.9 [35.9 to 53.9]

4. Secondary Outcome: Global Rating of Change Score of 3+ or Higher (Minimum Clinically Important Change)
Description: The GROC will be administered to patients at the 6 months, one year and two year time points. The GROC questionnaire is a common, feasible, and useful method for assessing short term outcomes and overall changes in quality of life and is a valid measurement of change in patient status in a variety of pain populations. The GROC has a 15-point scale with a change of positive three points or higher (3+) demonstrating clinically significant improvement in a patient's perception of quality of life. Scores of -1 to -7 indicate negative perception of improvement (worsening of condition), a 0 indicates no change, and scores of +1 through +7 indicate a positive perceived improvement in the patients condition.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arthroscopic Surgery | Physical Therapy
Number analyzed (Participants) | 37 | 37
Participants | 16 | 15

5. Other Pre Specified Outcome: Self-Motivation Inventory
Description: The Self-Motivation Inventory is an outcome measure that was developed to determine level of motivation. The Self-Motivation Inventory is a 40-item tool that has been found to measure an individual's tendency to persevere independent of situational reinforcement. It has also been used to predict successful weight loss and may correlate with number of sessions attended in weight loss program [29]. This tool underwent refinement in 1980 with the original 60-item tool being tested in undergraduate male and females. Items correlating less than 0.30 were deleted. The final 40-item scale yielded an exceptionally high internal reliability (α = 0.91) suggesting that a unitary common concept is evident for the obtained factor structure. The tool is widely used and has been tested in weight loss and therapeutic exercise studies
Time Frame: Baseline
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes From Baseline Pain Catastrophizing Scale at 24 Months
Description: The PCS is a 13-item patient-report scale developed to measure the extent to which people catastrophize in response to pain. Each item is scored from 0 ('not at all') to 4 ('all the time'). The PCS is reported as a total score, with higher scores indicating greater catastrophizing, and is composed of three sub-scales: Rumination (four items; e.g. 'When I am in pain, I keep thinking about how badly I want the pain to stop'), Magnification (three items; e.g. 'When I am in pain, I become afraid that the pain will get worse'), and Helplessness (six items; e.g. 'When I am in pain, I feel I can't go on'). The PCS has been shown to have high levels of internal consistency and construct validity.
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Arthroscopic Surgery | Physical Therapy
All-Cause Mortality (participants affected / at risk) | 1/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 2/40 | 2/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arthroscopic Surgery (N=40) | Physical Therapy (N=40)
Surgical complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) — Heterotopic ossification or femur fracture

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No